CLINICAL TRIAL: NCT00768495
Title: Evaluation of the Success of Endovascular Peripheral Revascularization for the Treatment of Chronic Limb Ischemia by Measuring OxyHb and DeoxyHb Using a New Hyperspectral Imaging Device (OxyVu).
Brief Title: Hyperspectral Imaging Pre and Post Endovascular Intervention
Acronym: CLI-Pre/Post
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: HyperMed (Industry)
Collaborators: Cardiac, Vascular & Thoracic Surgery Associates, P.C. (CVTSA) (Unknown)
Responsible Party: Kevin Schomacker, HyperMed, Inc.
Other Study IDs: 2008-023
Record Dates: First submitted 2008-10-06; First posted 2008-10-08 (Estimated); Last update posted 2009-06-04 (Estimated); Status verified 2009-06

CONDITIONS: Chronic Limb Ischemia; Non-Healing Ulcers
Keywords: revascularization; claudication; hyperspectral; oxygenation; limb ischemia
MeSH Terms: conditions — Intermittent Claudication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- One Cohort

SUMMARY:
This trial will collect tissue oxygenation data via hyperspectral imaging before and after endovascular procedures.

DETAILED DESCRIPTION:
This will be a nonrandomized, nonblinded, prospective observational study to correlate the results obtained with the traditional measures of success of endovascular revascularization of peripheral arteries for the treatment of chronic limb ischemia; i.e., ABPI, PVR with oxyhemoglobin (OxyHb) and deoxyhemoglobin (DeoxyHb) measurements obtained with a new imaging device manufactured by HyperMed Inc (OxyVu) that uses hyperspectral technology.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with established diagnosis of lower limb ischemic based on their symptoms of claudication, rest pain, non-healing ulcers or gangrene and other vascular laboratory tests that are currently used to make this diagnosis and have been scheduled for endovascular revascularization.
2. Age group between 50-85
3. Gender - Male or Female
4. Race - all race and ethnicities

Exclusion Criteria:

1. Patients with known cardiac disease - new MI (within 3 months).
2. Patients with hypertension with the systolic BP >200 or diastolic BP>110 on the day of testing
3. Patients on supplemental O2 for chronic obstructive lung disease
4. Bed-ridden subjects - either due to chronic disability or neurological problems

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have chronic limb ischemia and present with the symptoms of claudication, rest pain or having minor non-healing ulcers or gangrene (Rutherford category 1 to 6) who also require percutaneous endovascular revascularization.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Schomacker, PhD, Study Director — HyperMed
Locations (1):
- Cardiac, Vascular & Thoracic Surgery Associates, Falls Church, Virginia, United States

REFERENCES:
- [Background] Ostchega Y, Paulose-Ram R, Dillon CF, Gu Q, Hughes JP. Prevalence of peripheral arterial disease and risk factors in persons aged 60 and older: data from the National Health and Nutrition Examination Survey 1999-2004. J Am Geriatr Soc. 2007 Apr;55(4):583-9. doi: 10.1111/j.1532-5415.2007.01123.x. PMID 17397438
- [Background] White C. Clinical practice. Intermittent claudication. N Engl J Med. 2007 Mar 22;356(12):1241-50. doi: 10.1056/NEJMcp064483. No abstract available. PMID 17377162
- [Background] Yao ST. Haemodynamic studies in peripheral arterial disease. Br J Surg. 1970 Oct;57(10):761-6. doi: 10.1002/bjs.1800571016. No abstract available. PMID 5476754
- [Background] Begelman SM, Jaff MR. Noninvasive diagnostic strategies for peripheral arterial disease. Cleve Clin J Med. 2006 Oct;73 Suppl 4:S22-9. doi: 10.3949/ccjm.73.suppl_4.s22. PMID 17385388
- [Background] Raines JK, Darling RC, Buth J, Brewster DC, Austen WG. Vascular laboratory criteria for the management of peripheral vascular disease of the lower extremities. Surgery. 1976 Jan;79(1):21-9. PMID 1246689
- See also: Sponsor and OxyVu technology website — http://www.hypermed-inc.com